CLINICAL TRIAL: NCT06260943
Title: Targeted Navigation to Achieve Health Equity: Increasing Access to Care, Patient Engagement and Research Participation
Brief Title: Targeted Navigation in Hepatocellular Carcinoma (HCC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The V Foundation (Other)
Responsible Party: Principal Investigator, Patricia Jones, MD, Associate Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20221220; NCI-2024-00566 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Hepatobiliary Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aim 3: Targeted Navigation Pilot Program (Experimental): Participants in this group will be enrolled in a Targeted Navigation Pilot Program for up to 12 months.
  Interventions: Behavioral: Target Navigation Pilot Program

INTERVENTIONS:
Behavioral: Target Navigation Pilot Program — Participants will meet with a navigator, in either English, Spanish or Creole, biweekly, in person or virtually, until the first treatment appointment and every three months after. Each session will last approximately one hour; depending on the needs identified, patients will be connected to appropriate institutional or community-based resources.

SUMMARY:
The investigators are trying to learn more about the personal perceptions and experiences regarding the needs of patients with liver cancer to help improve the care of all patients. The investigators would like to know whether there are needs that patients have or are aware of, especially those needs that the investigators have not been able to address. The investigators aim to develop a program that helps participants and participant's families to navigate the process of being diagnosed with liver cancer and receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCC Patients:

  * Enrolled or eligible for enrollment in Unified Prospective Registry and Biorepository of Patients with Chronic Liver Disease or Hepatobiliary Cancers Including Hepatocellular Carcinoma (HCC) and Cholangiocarcinoma.
  * Diagnosis of hepatocellular carcinoma, confirmed by clinical chart review and International Classification of Diseases, Tenth Revision (ICD-10) C22.0.
  * Adults, age 18 or older
  * Able to provide informed consent
* All other interviewees:

  * Advocates who will self-identify as having had HCC.
  * Others who self-identify as either a caregiver or support person of an HCC patient.

Physicians/Licensed Independent Practitioners, Social Workers, Nurse Navigators, and Research Coordinators will all self-identify as being involved in the care of HCC patients.

Exclusion Criteria:

* Unable to speak Spanish or English
* West Haven Grade 2 or higher hepatic encephalopathy19 or other cognitive impairment.
* Adults unable or unwilling to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Given that this study is minimal risk and there are no risks to a potential fetus, investigators will not exclude pregnant women; however, no data about pregnancy or their fetus is being collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Days to First Contact | Up to 12 months
  The time to first contact since hepatocellular carcinoma diagnosis will be assessed in number of days.
Number of Hours for Each Contact | Up to 12 months
  The length of time of each contact will be assessed in number of hours. Contact is defined as the length of time the navigator meets with the participant.
Number of Days to First Appointment | Up to 12 months
  The time to first appointment will be assessed in number of days.
Number of Days to First Treatment | Up to 12 months
  The time to first treatment will be assessed in number of days.
Number of Months of Total Navigation | Up to 12 months
  The length of total navigation will be assessed in number of months.
Number of Participants that Die Within One Year | Up to 1 year
  Number of participants that die within one year of enrollment in the navigation program.
Proportion of Participants Enrolled in Clinical Research | Up to 12 months
  The proportion of participants enrolled in clinical research will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Jones, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No